CLINICAL TRIAL: NCT06674551
Title: Comparative Study Between Combined Suprascapular and Axillary Nerve Blocks Versus Interscalene Nerve Block Regarding Phrenic Nerve Affection Assessed by Ultrasound Guided Diaphragmatic Excursion in Shoulder Arthroscopy Surgeries
Brief Title: Suprascapular and Axillary Versus Interscalene Blocks Regarding Phrenic Affection in Shoulder Surgeries
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: FMASU MD128/2024
Record Dates: First submitted 2024-10-01; First posted 2024-11-05 (Actual); Last update posted 2024-11-05 (Actual); Status verified 2024-09

CONDITIONS: Interscalene Nerve Block; Suprascapular Nerve; Shoulder Surgery
Keywords: interscalene nerve block; axillary nerve block; shoulder surgery

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Suprascapular nerve block and Axillary nerve block ( Group A) (Experimental): Patients will receive Suprascapular nerve block (SSNB) and Axillary nerve block (AXNB) 30 minutes before the induction of general anaesthesia.
  Interventions: Procedure: Suprascapular nerve block and Axillary nerve block
- Interscalene nerve block (Group B) (Experimental): Patients will receive Interscalene nerve block (ISB) 30 minutes before the induction of general anaesthesia.
  Interventions: Procedure: Interscalene Nerve Block

INTERVENTIONS:
Procedure: Suprascapular nerve block and Axillary nerve block — A linear ultrasound probe will be placed in a sagittal plane at the superior medial border of the scapula. The probe will be moved laterally and then placed parallel to the scapular spine. when the needle tip contacts the bone just medial to the spinoglenoid notch and after confirmation of absence of vascular structure by color Doppler, 10 ml of 0.5% bupivacaine will be injected with aspiration every 3 ml to avoid intravascular injection and the spread of the local anaesthetic
  Arms: Suprascapular nerve block and Axillary nerve block ( Group A)
Procedure: Interscalene Nerve Block — The ultrasound probe will be placed in the supraclavicular fossa in a transverse orientation, aimed caudad into the thoracic cavity, to visualize the brachial plexus near the subclavian artery. Once identified, the plexus will be followed cephalad where it is found within the brachial plexus fascial sheath in the interscalene groove.
  Arms: Interscalene nerve block (Group B)

SUMMARY:
This study is aims to compare between combined suprascapular and axillary nerve blocks versus interscalene nerve block regarding phrenic nerve affection assessed by ultrasound guided diaphragmatic excursion in shoulder arthroscopy surgeries.

DETAILED DESCRIPTION:
Interscalene approach of brachial plexus nerve block is recognized as the gold standard technique for postoperative pain control after shoulder arthroscopy surgeries . However, it is associated with major adverse effects and possibly critical complications including phrenic nerve affection. Combined suprascapular and axillary nerve blocks are considered to be a safe and effective alternative to interscalene nerve block for shoulder surgery. Futher studies had been done regarding postoperative analgesia after shoulder arthroscopy surgeries using intersalene nerve block versus suprascapular and axillary nerve blocks.

In this study, we will Compare between combined suprascapular and axillary nerve blocks vs interscalene nerve block regarding objective phrenic nerve affection known as a serious complication of interscalene nerve block.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged between 18 - 60 years old.
* Both sexes.
* ASA physical status classes I - II.
* Body mass index: 18-35 kg/ m2.

Exclusion Criteria:

* Infection at site of injection.
* Psychiatric illness.
* Central Nervous System Diseases like (epilepsy, stroke …etc.) or neurological disease affecting patient's upper limb.
* Dependence on opiates and psycho-dynamic medications.
* Moderate to severe pulmonary disease.
* Coagulopathy and bleeding disorders.
* Allergies to drug used (Bupivacaine 0.5%).
* Previous surgery at site of injection and history of radiotherapy.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-11-20 (Estimated); Primary Completion 2025-10-01 (Estimated); Study Completion 2025-11-01 (Estimated)

PRIMARY OUTCOMES:
incidence of hemidiaphragmatic paralysis measured by ultrasound. | measurement will be taken 8 hours after the performance of the block for fourth and last time.
  defined as a ≥ 25% reduction in diaphragmatic excursion measured by ultrasound.

SECONDARY OUTCOMES:
postoperative pain using NRS | 24 hours postoperative
  is to measure first rescue analgesia postoperative (24 hours)